CLINICAL TRIAL: NCT05826886
Title: Social Learning in Depression Therapy: The Effect of Video-based Testimonials About Psychotherapy on a Treatment Expectations and a Short Online Intervention
Brief Title: The Effect of Video-based Testimonials About Psychotherapy on Treatment Expectations and a Short Online Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Winfried Rief, Professor, Dr., Philipps University Marburg
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: Social learning 2_intervention
Record Dates: First submitted 2023-03-22; First posted 2023-04-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Health Care Utilization
Keywords: treatment expectations; social learning; psychotherapy; depression; testimonials
MeSH Terms: conditions — Patient Acceptance of Health Care; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control video (Active Comparator): Video of a woman describing basic information about psychotherapy and how it is embedded in the insurance system in Germany. Personal experience with therapy are not provided. 'Emotional writing' is introduced as a type of intervention used in depression treatment and basic information about it is provided.
  Interventions: Behavioral: Emotional Writing
- Testimonials (Experimental): Video of a patient and a therapist, who both describe their personal experience of depression therapy in a positive but realistic way. Emphasis is on the personal experience protagonist. 'Emotional writing' is described as a helpful technique from a first person perspective.
  Interventions: Behavioral: Emotional Writing

INTERVENTIONS:
Behavioral: Emotional Writing — Participants complete four 20-minute sessions of emotional writing (at home) on four consecutive days. Instructions are provided online before each writing session.
  Other Names: Expressive Writing

SUMMARY:
Research has shown that treatment expectations play a major role in the course of mental disorders and that positive expectations have a beneficial impact on treatment outcomes. Expectations can develop in different ways and an emerging body of research shows that social learning plays a significant role in this process. To date, most studies have investigated the impact of social learning on treatment expectations in the context of pain relief. Little is known about the impact of social learning in the psychotherapeutic treatment of depression. Therefore, this study investigates whether treatment expectations about depression therapy and treatment effects of a short online intervention can be modulated via social learning, i.e., showing positive treatment testimonials.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* be able understand German (at least B1 level)
* have access to a computer device with internet access

Exclusion Criteria:

* age below 18 years old
* non correctable hearing or visual impairment
* diagnosis of borderline-personality disorder
* diagnosis of post-traumatic-stress-disorder
* self-reported suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in scores on the Credibility and Expectancy Questionnaire (CEQ) scale | Baseline; after viewing the videos (1 day after baseline); after completion of the writing intervention (5 days after baseline)
  German version of the Credibility and Expectancy Questionnaire (CEQ), 6-item scale.The CEQ consists of two subscales with four items measuring cognitive-focused credibility (e.g., "At this point, how logical does the therapy offered to you seem?") and two items measuring affect-focused expectations (e.g., "By the end of the therapy period, how much improvement in your symptoms do you really feel will occur?"). The CEQ applies different rating scales; a 9-point scale ranging from 1 (not at all) to 9 (very much) and a percentage rating scale ranging from 0% (not at all) to 100% (very much) with higher sum scores indicating greater treatment credibility and expectations.
Change from baseline in scores on self-report measure for the Assessment of Emotion Regulation Skills (Fragebogen zur standardisierten Selbsteinschätzung emotionaler Kompetenzen; SEK-27) | Baseline; after completion of the writing intervention (5 days after baseline)
  The German SEK-27 is a 27-item scale measuring 9 domains (attention, clarity, body awareness, understanding, acceptance, resilience, self-support, readiness for confrontation, and regulation) of emotion regulation skills. Higher scores on the overall score indicate better emotion regulation skills.

SECONDARY OUTCOMES:
Change from baseline in scores on the Patient Health Questionnaire (PHQ-9) | Baseline; after completion of the writing intervention (5 days after baseline)
  Depressive symptoms via the German version of the Patient Health Questionnaire (PHQ-9), 9-item scale. With each item, the PHQ-9 captures one of the nine criteria for major depression posted in the Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) using a 4-point Likert-scale ranging from 0 (not at all) to 3 (almost every day). The total score ranges of 0 to 27, whereby a score of 0 to 4 indicates minimal depressive symptomatology, a score of 5 to 9 mild, a score of 10 to 14 moderate, a score of 15 to 19 moderate to severe, and a total score of 20 to 27 severe depressive symptomatology.
Change from baseline in subjective stress scores on the 'Perceived Stress Scale' (PSS-10) | Baseline; after completion of the writing intervention (5 days after baseline)
  Self-report questionnaire to assess subjective stress experience; 10 items; each item is rated on a 5-point scale from 0(never) to 4(very often); total scores range between 0 and 40 (higher scores indicate more subjective stress).
Change from baseline in scores on Regulatory Emotional Self-Efficacy Scale (RESE) | Baseline; after completion of the writing intervention (5 days after baseline)
  The German version of the RESE is a 10-item instrument measuring self-efficacy for emotion regulation. Items are scored on a Likert Scale ranging from 1 (not well at all) to 5 (very well). Higher scores indicate better regulatory emotional self-efficacy.
Change from baseline on the state-anxiety subscale of the 'State-Trait-Anxiety- Depression-Inventory' (STADI) | Baseline; after completion of the writing intervention (5 days after baseline)
  Self-report questionnaire to assess state and trait anxiety and depression; 40 (20 state scale; 20 trait scale) items; each item is rated on a 4-point scale from 1(not at all) to 4(very much); total scores per scale range between 20 and 80 (higher scores indicate more anxiety)
Change from baseline in scores on specific emotion regulation items | Baseline; after completion of the writing intervention (5 days after baseline)
  Because we felt that the existing emotion regulation scales used in this study did not capture the some of the specific skills that the emotional writing intervention targets, we created a set of five specific items about allowing, accepting, experiencing and managing negative emotions. Items are scored on a Likert Scale ranging from 1 (do not agree at all) to 5 (agree completely). Higher scores indicate better emotion regulation abilities.
Change from baseline in scores on the treatment expectations subscale of the the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE) | Baseline; after viewing the videos (1 day after baseline); after completion of the writing intervention (5 days after baseline)
  Treatment expectations are measured via the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE), subscale for previous treatment experiences and subscale for treatment expectations. Answers are provided on a numeric rating scale ranging from 0 to 10 (each item has specific anchors with lower anchors always indicating no expected effects)
Change from baseline in scores on perceived uncertainty and perceived barriers to psychotherapy | Baseline; after viewing the videos (1 day after baseline)
  The items used by Kushner and Sher (1989), to assess perceived barriers were translated to German and modified to state "I am uncertain" instead of "I am anxious". The scale consists of 3 subscales: therapist responsiveness (5 items), image concerns (4 items), coercion concerns (4 items). Answers are provided on a 5-point scale ranging from 1 (not at all) to 5 (completely) with high scores indicating greater uncertainty. Five items to reflect specific uncertainties (financial concerns, time restrictions, therapist relatability, the therapeutic process, personal ability to complete therapy), that were not covered by the original article, were added. Answers are provided on a 5-point scale ranging from 1 (do not agree) to 5 (agree) with high scores indicating greater uncertainty.
Change from baseline in scores on the Credibility and Personal Reaction Scale | Baseline; after viewing the videos (1 day after baseline); after completion of the writing intervention (5 days after baseline)
  Credibility of and personal reactions to psychotherapy are measured via a self-translated German version of the Credibility & Personal Reaction Scale. This scale also measures intentions to seek therapy.
  Credibility scale: 7 items, answers are provided on a 7-point Likert scale from 1 (not at all) to 7 (extremely).
  Personal Reactions to the Rationales (PRR): 5 items, answers are provided on a 7-point Likert scale from 1 (not at all) to 7 (extremely).
  The total score of the credibility scale ranges from 7 to 49 with higher scores indicating higher credibility ratings, the total PRR score ranges from 5 to 35 with higher scores indicating more positive reactions and higher credibility.
Change from baseline in D-Scores on the Single-Category Implicit Associations Test (SC-IAT) | Baseline; after viewing the videos (1 day after baseline)
  Single-Category Implicit Associations Test (SC-IAT), measuring implicit associations with psychotherapy. It is a reaction-time task facing the target dimension 'psychotherapy' and the evaluative dimensions 'effective' and 'ineffective'. The strength of the association (D-score) between the target dimension and the evaluative dimension is calculated based on the reaction times. Shorter reaction times indicate a greater associative strength.
Change from baseline in scores on the Self-Stigma of Depressions Scale (SSDS) | Baseline; after viewing the videos (1 day after baseline)
  German version of the Self-Stigma of Depressions Scale (SSDS), 16 items measuring anticipated self-stigma for the hypothetical case that one would be suffering from depression. The SSDS consists of 3 subscales: self-blame, help-seeking inhibition, social inadequacy Answers on all items are given on a 5-point Likert-scale ranging from 1 (completely disagree) to 5 (completely agree); higher scores indicate higher self-stigma.
Change from baseline in the items assessing expectations about dealing with negative emotions of the Depressive Expectations Scale (DES) | Baseline; after completion of the writing intervention (5 days after baseline)
  Part A (6 items) of the Depressive Expectations Scale (DES). Items are scored on a Likert Scale ranging from 1 (do not agree) to 5 (agree). Higher scores indicate stronger negative expectations about dealing with negative emotions.

OTHER OUTCOMES:
General Self-Efficacy Scale (GSE) | Baseline
  Self-efficacy via the German version of the General Self-Efficacy Scale (GSE), a 10-item scale measuring general self-efficacy. The scale contains 10 items (e.g., "When I am confronted with a problem, I can usually find several solutions"). The answers are presented on a 4-point Likert-scale ranging from 1 (not true at all) to 4 (exactly true) which yields a total score between 10 and 40 with high scores indicating high levels of general self efficacy perceptions.
Locus of control perceptions/ "Internale-Externale-Kontrollüberzeugungen-4" (IE-4) | Baseline
  The German 4-item scale Internale-Externale-Kontrollüberzeugungen-4 (IE-4) to assess locus of control.
  The IE-4 scale consists of 2 subscales: internal (2 items) and external locus of control (2 items). The 4 items are answered using a 5-point Likert-scale ranging from 1 (strongly disagree) to 5 (strongly agree). The subscale scores are averaged into one score per subscale. The mean subscale values range between 1 and 5 with higher scores indicating higher internal or external locus of control.
Empathy on the Interpersonal Reactivity Index (IRI) | Baseline
  Empathy via the German version of the Interpersonal Reactivity Index (IRI), a 16-item scale. Answers are provided on a 5-point rating scale ranging from 1 (never) to 5 (always). Empathy is divided into one cognitive and three emotional components: perspective taking (PT; item 4,10,14,16), fantasy scale (FS; item 2,7,12,15), empathic concern (EC; 1,5,9,11) and personal distress (PD; 3,6,8,13); the general score is determined by the sum value of the individual scales EC, PT and FS (empathy=EC+PT+FS), whereby a higher score indicates higher empathy.
Cognitive Emotion Regulation Questionnaire (CERQ) | Baseline
  The CERQ-short is an 18-item instrument measuring the habitual use of adaptive and maladaptive cognitive emotion regulation styles (self-blame, rumination, acceptance, positive refocusing, refocus on planning, positive reappraisal, putting into perspective, catastrophizing, other-blame) with 2 items per subscale. Items are scored on a Likert Scale ranging from 1 (almost never) to 5 (almost always). Higher scores indicate more frequent use of a cognitive emotion regulation style.
Perceived Stigma subscale of the Depression Stigma Scale (DSS) | Baseline
  Public Stigma of depression are measured via the German translation of the Depression Stigma Scale (DSS), using the Perceived Stigma subscale: 9 items, measuring perceived public stigma of depression. Answers are provided on a 5-point Likert-scale ranging from 0 (completely disagree) to 4 (completely agree); total scores range from 0 to 36 with higher scores indicating greater perceived stigma.
Previous treatment experiences on the subscale for previous treatment experiences of the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE) | Baseline
  Prior experiences with psychotherapy are measured via the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE), subscale for previous treatment experiences. Answers are provided on a numeric rating scale ranging from 0 to 10 (each item has specific anchors with lower anchors always indicating no expected effects)
Cognitive Immunization (of the video information) | after completion of the writing intervention (5 days after baseline)
  Four items to assess tendencies to discredit the information viewed in the intervention videos.
Process questions about the intervention | at every emotional writing session (1 day, 2 days, 3 days, 4 days after baseline)
  We created three items relating to dealing with emotions before, after and during the emotional writing session. The three items assess: mood in the past 24 hours (item scored on a 10-point Likert Scale; higher scores indicate better mood), ability to cope with emotions in the past 24 hours (item scored on a 10-point Likert Scale; higher scores indicate more ability to cope with emotions), adherence to the emotional writing session (item scored on a 10-point Likert Scale; higher scores indicate more adherence). A forth item was taken from the Depressive Expectations Scale (DES) to assess the expectation about the ability to cope with emotions in the coming 24 hours (item scored on a Likert Scale ranging from 1 (do not agree) to 5 (agree). Higher scores indicate stronger negative expectations about coping with negative emotions in the next 24 hours)
Current treatment effects subscale of the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE) | after completion of the writing intervention (5 days after baseline)
  Current treatment effects are measured via the current treatment effects subscale of the generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE). Answers are provided on a numeric rating scale ranging from 0 to 10 (each item has specific anchors with lower anchors always indicating no expected effects)
Warmth and competence ratings of the actors shown in the videos | after viewing the videos (1 day after baseline, directly after viewing the intervention videos)
  Participant perceptions of warmth and competence of actors shown in the videos are measured via the Warmth and Credibility Screener - German translation: 12 items assessing perceived warmth (6 items) and competence (6 items) on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely) with high scores indicating greater ratings of warmth and competence.

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Principal Investigator — Department of Clinical Psychology and Psychotherapy, Philipps-University Marburg, Germany
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Philipps-University Marburg, Marburg, Germany

REFERENCES:
- [Background] Koch SC, Mergheim K, Raeke J, Machado CB, Riegner E, Nolden J, Diermayr G, von Moreau D, Hillecke TK. The Embodied Self in Parkinson's Disease: Feasibility of a Single Tango Intervention for Assessing Changes in Psychological Health Outcomes and Aesthetic Experience. Front Neurosci. 2016 Jul 7;10:287. doi: 10.3389/fnins.2016.00287. eCollection 2016. PMID 27458332
- [Background] Berking, M., & Znoj, H. (2008). Entwicklung und Validierung eines Fragebogens zur standardisierten Selbsteinschätzung emotionaler Kompetenzen (SEK-27). Zeitschrift für Psychiatrie, Psychologie und Psychotherapie, 56(2), 141-153.
- [Background] Lowe B, Kroenke K, Herzog W, Grafe K. Measuring depression outcome with a brief self-report instrument: sensitivity to change of the Patient Health Questionnaire (PHQ-9). J Affect Disord. 2004 Jul;81(1):61-6. doi: 10.1016/S0165-0327(03)00198-8. PMID 15183601
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Gunzenhauser, C., Heikamp, T., Gerbino, M., Alessandri, G., Von Suchodoletz, A., Di Giunta, L., ... & Trommsdorff, G. (2013). Self-efficacy in regulating positive and negative emotions. European Journal of Psychological Assessment, 29(3):197-204.
- [Background] Renner KH, Hock M, Bergner-Kother R, Laux L. Differentiating anxiety and depression: the State-Trait Anxiety-Depression Inventory. Cogn Emot. 2018 Nov;32(7):1409-1423. doi: 10.1080/02699931.2016.1266306. Epub 2016 Dec 8. PMID 27928931
- [Background] Rief, W., Nestoriuc, Y., Mueller, E. M., Hermann, C., Schmidt, K., & Bingel, U. (2021). Generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE). PsychArchives. https://doi.org/10.23668/PSYCHARCHIVES.4717
- [Background] Kushner, M. G., & Sher, K. J. (1989). Fear of psychological treatment and its relation to mental health service avoidance. Professional Psychology: Research and Practice, 20(4), 251.
- [Background] Addis ME, Carpenter KM. Why, why, why?: Reason-giving and rumination as predictors of response to activation- and insight-oriented treatment rationales. J Clin Psychol. 1999 Jul;55(7):881-94. doi: 10.1002/(sici)1097-4679(199907)55:73.0.co;2-e. PMID 10866023
- [Background] Karpinski A, Steinman RB. The single category implicit association test as a measure of implicit social cognition. J Pers Soc Psychol. 2006 Jul;91(1):16-32. doi: 10.1037/0022-3514.91.1.16. PMID 16834477
- [Background] Makowski AC, Mnich EE, von dem Knesebeck O. [Self-Stigma of Depression Scale SSDS - Evaluation of the German Version]. Psychiatr Prax. 2018 Sep;45(6):314-320. doi: 10.1055/s-0043-104504. Epub 2017 May 12. German. PMID 28499317
- [Background] Kube T, D'Astolfo L, Glombiewski JA, Doering BK, Rief W. Focusing on situation-specific expectations in major depression as basis for behavioural experiments - Development of the Depressive Expectations Scale. Psychol Psychother. 2017 Sep;90(3):336-352. doi: 10.1111/papt.12114. Epub 2016 Dec 9. PMID 27935247
- [Background] Kovaleva, A., Beierlein, C., Kemper, C. J., & Rammstedt, B. (2012). Eine Kurzskala zur Messung von Kontrollüberzeugung: die Skala Internale-Externale-Kontrollüberzeugung-4 (IE-4). (GESIS-Working Papers, 2012/19). Mannheim: GESIS - Leibniz-Institut für Sozialwissenschaften. https://nbn-resolving.org/urn:nbn:de:0168-ssoar-312096
- [Background] Paulus, C. (2009). DER SAARBRÜCKER PERSÖNLICHKEITSFRAGEBOGEN SPF(IRI) ZUR MESSUNG VON EMPATHIE: Psychometrische Evaluation der deutschen Version des Interpersonal Reactivity Index. https://doi.org/10.23668/psycharchives.9249
- [Background] Garnefski, N., & Kraaij, V. (2006). Cognitive emotion regulation questionnaire-development of a short 18-item version (CERQ-short). Personality and individual differences, 41(6), 1045-1053.
- [Background] Griffiths KM, Christensen H, Jorm AF. Predictors of depression stigma. BMC Psychiatry. 2008 Apr 18;8:25. doi: 10.1186/1471-244X-8-25. PMID 18423003
- [Background] Seewald, A., & Rief, W. (2023). How to change negative outcome expectations in psychotherapy? The role of the therapist's warmth and competence. Clinical Psychological Science, 11(1), 149-163.